CLINICAL TRIAL: NCT04430595
Title: Multiple 4SCAR-T Cell Therapy Targeting Breast Cancer
Brief Title: Multi-4SCAR-T Therapy Targeting Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20005
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: CART; adoptive T cell transfer; Her2; GD2; CD44V6
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple 4SCAR T cells to treat breast cancer (Experimental): Multiple 4SCAR T cells to treat breast cancer
  Interventions: Biological: 4SCAR T cells

INTERVENTIONS:
Biological: 4SCAR T cells — Infusion of 4SCAR-GD2, -Her2 and -CD44v6 CAR-T cells

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of multiple 4th generation CAR-T cells targeting Her2, GD2, and CD44v6 surface antigen in breast cancer. Another goal of the study is to learn more about the activities of the multi-CAR T cells and their persistency in the patients.

DETAILED DESCRIPTION:
Breast cancer is one of the most frequent cancer types in women. The average risk of a woman in the United States developing breast cancer in her life is about 13%. That means that there is a 1 in 8 chance she will develop breast cancer. Human epidermal growth factor receptor-2 (HER2) is one of the more well-researched genes in breast cancer so far. It has been reported that HER2 gene is overexpressed in 20% to 30% of breast cancer patients. HER2 is an important target for tumor gene therapy. In 2003, scientists confirmed the existence of breast cancer stem cells. In 2012, ganglioside GD2 was confirmed as an emerging marker of breast cancer stem cells. Targeting therapies for GD2 may help improve the survival rate and cure rate of breast cancer patients. Invasion and metastasis of tumor cells is the main cause of cancer death. CD44v6 is an adhesion molecule on the cell surface, which not only promotes epithelial-mesenchymal transition, degradation and remodeling of extracellular matrix, but also participates in organ-specific metastasis of tumor cells. Studies have shown that overexpression of CD44v6 is an important factor for the invasion and metastasis of breast cancer, and is closely related to the tumor size of the breast cancer, tumor staging, and lymph node metastasis. Therefore, CD44v6 may be an important target for the treatment of breast cancer. Using Her2-, GD2- and CD44v6-specific CAR-T cells may effectively improve the immunotherapy treatment, prevent tumor cells from escaping treatment, and achieve the effect of long-term disease relief.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III, IV or relapsed breast cancer confirmed by histology and biopsy.
2. Age: ≥ 18 years and ≤ 75 years.
3. 2 weeks at least since last chemotherapy or radiotherapy and 2 weeks at least since last systemic steroid hormone and other immunosuppressive therapy.
4. Side effects of chemotherapy have subsided.
5. The target antigens GD2, CD44v6, or Her2 is expressed in malignancy tissues by immuno-histochemical or flow cytometry.
6. Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
7. Expected survival ≥ 12 weeks.
8. Initial hematopoietic reconstitution with neutrophils (ANC) ≥ 1×10^6/L; platelet (PLT) ≥ 1×10^8/L.
9. Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with serum creatinine ≤ 2×ULN; serum bilirubin ≤ 3×ULN; AST/ALT ≤ 2.5×ULN.
10. Oxygen saturation ≥ 90%.
11. Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

1. Airway obstruction caused by tumor.
2. History of epilepsy or other central nervous system diseases.
3. Patients who require systemic corticosteroid or other immunosuppressive therapy.
4. History of prolonged or serious heart disease during QT.
5. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug or previous participation in this study.
6. Inadequate liver and renal function with serum creatinine > 1.5 mg/dl; serum (total) bilirubin > 2.0 mg/dl; AST & ALT > 3 x ULN.
7. Pregnant or lactating females.
8. Serious active infection during screening.
9. Active HIV, hepatitis B virus (HBV), hepatitis C virus (HCV) infection or uncontrolled infection.
10. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 3 year
  Determine the toxicity profile the multi-4SCAR-T cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 3 year
  Disease status is defined by the image scan to get the outcomes such as Complete response/remission (CR), Very good partial response/remission (VGPR), etc.
The expansion and persistence of CAR-T cells | 3 months
  The expansion and functional persistence of CART cells in the peripheral blood of patients will be measured by qPCR on Day 7, 14, 21, 28, 60 and 90 after infusion.
Survival time of the patients | 3 year
  The survival time of the patients treated with the multi-4SCAR T cells, including progression free survival (PFS) and overall survival (OS) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- The Seventh Affilliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No